CLINICAL TRIAL: NCT03215823
Title: Predictive Factors of the Difficult Intubation When Using the Videolaryngoscope
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 1-2017-0035
Record Dates: First submitted 2017-07-09; First posted 2017-07-12 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Endotracheal Intubation Using Videolaryngoscope for General Anesthesia
Keywords: Intubation; videolaryngoscope

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1. Easy endotracheal intubation: Easy endotracheal intubation
- 2. Difficult endotracheal intubation: Difficult endotracheal intubation

SUMMARY:
The usefulness of videolaryngoscope has been verified by several studies, and the frequency of videolaryngoscopy is increasing in clinical practice. Data on the use of videolaryngoscopes, however, were not sufficiently accumulated when compared with data on the use of previously used macintosh laryngoscopes. In addition, videolaryngoscopy increases the success rate of endotracheal intubation compared to conventional macintosh laryngoscopy, but endotracheal intubation with videolaryngoscope is not successful in all cases with one intubation attempt. Therefore, if the difficult endotracheal intubation with the videolaryngoscope can be predicted in advance, it may be possible to improve the success rate of intubation by reducing unnecessary use of the videolaryngoscope and preparing other equipment. There are many studies on the preoperative examination that can predict the difficulty of intubation when using a macintosh laryngoscope. However, there are still attempts to find screening tests that predict precisely the difficult endotracheal intubation because the accuracy of screening tests is not high. In particular, there is a lack of research on factors that can predict difficult endotracheal intubation when using videolaryngoscope. Therefore, the investigators aimed to investigate the factors predictive of difficult endotracheal intubation when attempting intubation using videolaryngoscope.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are scheduled for endotracheal intubation using a videolaryngoscope for general anesthesia

Exclusion Criteria:

1. Patients who are planned to receive awake intubation
2. Patients who have a tracheostomy tube
3. Patients who do not cooperate in evaluating the head and neck due to mental retardation
4. Trauma patient wearing a neck collar due to cervical fracture
5. Pregnancy

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are scheduled for endotracheal intubation using videolaryngoscope for general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 808 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2018-11-14 (Actual); Study Completion 2018-11-14 (Actual)

PRIMARY OUTCOMES:
the occurrence of the difficult endotracheal intubation when using a videolaryngoscope. | 10 minutes during the induction of general anesthesia.
  logistic regression analysis will be used to find out the predictors of the difficult endotracheal intubation.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Stoneham MD. The nasopharyngeal airway. Assessment of position by fibreoptic laryngoscopy. Anaesthesia. 1993 Jul;48(7):575-80. doi: 10.1111/j.1365-2044.1993.tb07119.x. PMID 8346770
- [Result] Reed DB, Clinton JE. Proper depth of placement of nasotracheal tubes in adults prior to radiographic confirmation. Acad Emerg Med. 1997 Dec;4(12):1111-4. doi: 10.1111/j.1553-2712.1997.tb03691.x. PMID 9408424
- [Result] Han DW, Shim YH, Shin CS, Lee YW, Lee JS, Ahn SW. Estimation of the length of the nares-vocal cord. Anesth Analg. 2005 May;100(5):1533-1535. doi: 10.1213/01.ANE.0000149900.68354.33. PMID 15845720
- [Derived] Kim HJ, Kim HR, Kim SY, Kim HY, Park WK, Lee MH, Kim HJ. Predictors of difficult intubation when using a videolaryngoscope with an intermediate-angled blade during the first attempt: a prospective observational study. J Clin Monit Comput. 2022 Aug;36(4):1121-1130. doi: 10.1007/s10877-021-00742-9. Epub 2021 Jul 12. PMID 34251587